CLINICAL TRIAL: NCT03496129
Title: Evaluation of an Interactive Text-Message Based Brief Intervention to Reduce Substance-Impaired Driving Among College Students
Brief Title: An Interactive Text-Message Based Brief Intervention to Reduce Substance-Impaired Driving Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-187
Record Dates: First submitted 2018-04-03; First posted 2018-04-12 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alcohol-Impaired Driving

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Feedback (Experimental): Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback. Feedback will include the following elements: a personalized substance use profile and substance-impaired driving profile, information on social norms related to substance use and substance-impaired driving, personalized information on BAC (or level of impairment due to drug use) prior to driving, costs associated with a DUI citation in Kentucky, and information on combined drug and alcohol impaired driving risk (if endorsed).
  Interventions: Behavioral: Personalized feedback
- Personalized feedback and text messages (Experimental): Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
  Interventions: Behavioral: Personalized feedback and text messages
- Information Only (Active Comparator): Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
  Interventions: Behavioral: Information Only

INTERVENTIONS:
Behavioral: Personalized feedback — Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback. Feedback will include the following elements: a personalized substance use profile and substance-impaired driving profile, information on social norms related to substance use and substance-impaired driving, personalized information on BAC (or level of impairment due to drug use) prior to driving, costs associated with a DUI citation in Kentucky, and information on combined drug and alcohol impaired driving risk (if endorsed).
  Arms: Personalized Feedback
Behavioral: Personalized feedback and text messages — Experimental: Personalized feedback and text messages
  Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
  Arms: Personalized feedback and text messages
Behavioral: Information Only — Active Comparator: Information Only
  Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
  Arms: Information Only

SUMMARY:
Substance-Impaired Driving among college students remains a significant public health concern and may be the single riskiest substance-related outcome among young adults. Brief Interventions (BIs) have been shown to reduce alcohol-impaired driving among college students, but are not often implemented - despite their demonstrated efficacy - because it is not economically feasible for universities to hire and train staff to deliver in-person BIs to all college substance users. Very few college students seek out substance prevention or treatment services available on campus or in the surrounding community. Innovative ways of delivering BIs to this at-risk population in a manner that is both effective and economically feasible have to be developed. The present study will be the first to examine whether a text-messaging-based substance-impaired driving BI significantly decreases substance-impaired driving among colleges substance users compared to an informational control. Participants will be 150 college students who endorse driving after substance use (alcohol, drugs, and/or combined alcohol/drugs) at least twice in the past 3 months. After completing baseline measures, participants will be randomly assigned to receive either: a) substance use information, b) a substance-impaired driving personalized feedback intervention, or c) a substance-impaired driving personalized feedback intervention plus interactive text messages. Participants will complete outcome measures 3, 6, and 12 months post-intervention. Repeated measures mixed modeling analyses will be used to determine whether the intervention significantly reduces substance-impaired driving over time. The project has two specific aims: 1) to evaluate a text based substance-impaired driving intervention in a randomized clinical trial, and 2) to determine whether the use of interactive text-messages sustains intervention effects over time. This study is innovative because it utilizes cutting-edge technology to deliver the entire intervention, enabling the study to reach a large number of students in a short time period at a low cost. The study is significant because it will contribute substantially to the substance-impaired driving literature by identifying an intervention that can decrease substance-impaired driving among this high-risk population. Additionally, this study will add to the newly emerging technology-based intervention literature.

DETAILED DESCRIPTION:
Rates of substance-impaired driving remain especially high among college students, and substance-related traffic accidents remain the leading cause of substance-related death among young adults. Prevention and intervention efforts, such as brief Interventions (BIs) have been shown to decrease substance use and related problems. BIs attempt to identify and correct faulty normative beliefs and highlight consequences of substance use (such as driving after substance use) and BIs typically consist of one or two individual therapeutic meetings delivered in motivational interviewing style and include personalized feedback (based on a series of questionnaires completed by the student prior to their BI session). The reason why BIs have not been deployed - despite their demonstrated efficacy - is that it is not economically feasible for universities to hire and train staff to deliver in-person BIs to all college substance users, and very few college students seek out substance prevention or treatment services available on campus or in the surrounding communities. Innovative ways of delivering BIs to this at-risk population in a manner that is both effective and economically feasible have to be developed. Text messaging represents a particularly advantageous way to provide BIs as they can be highly personalized to the individual, accessed at any time that suits the individual's needs, and allow for engagement and interaction between the interventionist and participant. Given the high prevalence and fatal consequences of substance-impaired driving, intervention approaches with the ability to reach a large number of students at a low cost are imperative for reducing this extremely risky behavior. Personalized feedback delivered without a one-on-one intervention may effectively reduce substance use and problems, despite the fact that web-based and feedback-only interventions consistently demonstrate smaller effect sizes than in-person interventions at long-term follow-ups, with effects often dissipating after the first follow-up.

The present study will enhance and extend intervention effects by including MI consistent interactive text messages to provide an interpersonal and interactive element. Research indicates that college students prefer text messages to telephone calls and emails and rate this medium positively. However, few published studies in alcohol literature have implemented text-messaging interventions and no published studies have examined the effects of a text-based substance impaired driving BI among students who report recent substance-impaired driving. A text-based BI focused specifically on decreasing alcohol-impaired driving (AI-driving) among college students has been developed and evaluated in a pilot trial. This study indicated that a brief, text-based AI-driving intervention resulted in significantly greater reductions in AI-driving at the 3-month follow-up, compared to an intervention providing alcohol information alone. This was the first controlled study to demonstrate that a text-based AI-driving intervention could decrease AI-driving outcomes over time. However, it is not clear from this study whether interactive text messages are a crucial part of the intervention because this study did not compare an AI-driving feedback only condition to the AI-driving feedback + interactive texts condition.

The proposed study will extend these promising pilot results by (a) expanding inclusion criteria to include drug-impaired and combination drug and alcohol-impaired drivers, (b) increasing power and generalizability by recruiting 150 college students indicating recent substance-impaired driving, (c) dismantling the pilot trial design by including a personalized feedback only condition, and (d) including a 6-month and 1-year follow-up to determine whether intervention effects persist over time.

The overarching goal is to reduce driving after drinking, drug use, and combined drug/alcohol use among college students.

We will conduct a 3-group trial with 150 college students (project 50% female and 20% minority) recruited from a large public university.

Group 1: substance information only Group 2: substance-impaired driving personalized feedback only Group 3: substance impaired driving personalized feedback and MI interactive text messages

Aim 1: Evaluate a text based substance-impaired driving intervention in a Randomized Clinical Trial.

Hypothesis 1: Groups 2 and 3 will report greater reductions in driving after substance use at 3-month follow-up compared to Group 1.

Aim 2: Determine whether interactive text-messages sustain intervention effects over time.

Hypothesis 2: Group 3 will report greater reductions in driving after substance use at 6-month and 12-month follow-up compared to Group 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently enrolled (full or part-time) in college
* Ability to speak, read, and write in English
* Reports driving after drinking two or more drinks prior to driving at least three times in the past three months AND/OR reports driving after using marijuana or any other substance prior to driving at least three times in the past three months
* Reports having access to a motor vehicle, a valid driver's license, and plans to drive a vehicle in the next 3 months
* Reports access to a cell phone and willingness to read intervention material and exchange 3 texts post intervention with the study administrator
* Reports a valid email address

Exclusion Criteria:

* Currently in treatment for substance use or abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-09-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenni B Teeters, PhD, Principal Investigator — Western Kentucky University
Locations (1):
- Gary Ransdell Hall, Bowling Green, Kentucky, United States

REFERENCES:
- [Derived] Teeters JB, King SA, Hubbard SM. A mobile phone-based brief intervention with personalized feedback and interactive text messaging is associated with changes in driving after cannabis use cognitions in a proof-of-concept pilot trial. Exp Clin Psychopharmacol. 2021 Apr;29(2):203-209. doi: 10.1037/pha0000442. PMID 34043401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via flyers around campus, the Sona system, and a mass email sent out to all students.
Pre-assignment Details: Eight participants screened eligible and were randomized after completing their baseline survey per the study protocol. However, they were then deemed ineligible after reviewing their answers on the baseline survey. These participants were then taken out of the trial and not included in any data analyses.
Groups:
- Personalized Feedback and Text Messages: Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
  Personalized feedback and text messages: Experimental: Personalized feedback and text messages
  Following the baseline assessment, participants will be sent a link via text message to a secure website containing substance-impaired driving specific personalized feedback (described above). Participants will be asked to send a text message back to the study administrator after viewing the feedback document. After confirming receipt and processing of the document, the study administrator will then send the participant three text messages containing open-ended questions.
- Information Only: Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
  Information Only: Active Comparator: Information Only
  Students randomized to the information condition will receive standard information about alcohol and other drugs and substance-impaired driving via a link to a website delivered through text message.
Period: Overall Study
Arm/Group | Personalized Feedback | Personalized Feedback and Text Messages | Information Only
Started | 30 | 40 | 35
Completed | 28 | 38 | 31
Not Completed | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Per study protocol, participants who are eligible on the screening survey are randomized to one of three conditions.
Groups:
- Personalized Feedback: Received personalized feedback intervention.
- Personalized Feedback and Text Messages: Received personalize feedback and interactive text messages.
- Information: Received generic information about substance use and driving.
- Total: Total of all reporting groups
Arm/Group | Personalized Feedback | Personalized Feedback and Text Messages | Information | Total
Number analyzed (Participants) | 28 | 38 | 31 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 38 | 31 | 97
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 25 | 21 | 64
  Male | 10 | 10 | 9 | 29
  Non-binary | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 105 participants were randomized but only 97 completed all required study procedures and were included in data analyses.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Asian | 0 | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 3 | 4 | 7
    White | 25 | 27 | 26 | 78
    More than one race | 2 | 2 | 0 | 4
    Unknown or Not Reported | 0 | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 38 | 31 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Times Driving After Using Substances
Description: Participants will be asked to report the number of times they have driven within two hours of drinking alcohol or using other substances.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Driving Events
Arm/Group | Personalized Feedback | Personalized Feedback and Text Messages | Information Only
Number analyzed (Participants) | 28 | 38 | 31
Driving Events | 22.43 (21.39) | 26.50 (26.55) | 26.00 (25.46)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Personalized Feedback | Personalized Feedback and Text Messages | Information Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03496129/Prot_SAP_000.pdf